CLINICAL TRIAL: NCT01577628
Title: Randomized, Multicentric, Controlled Study on the Daily Use of Lipikar Balm AP From Birth in Infants at High Risk of Developing Atopic Dermatitis
Brief Title: Daily Use of Lipikar Balm AP From Birth in Infants at High Risk of Developing Atopic Dermatitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Cosmetique Active International (Industry)
Collaborators: Innovaderm Research Inc. (Other)
Responsible Party: Principal Investigator, Robert BISSONNETTE, President and Dematologist, Cosmetique Active International
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LRP11005
Record Dates: First submitted 2012-04-10; First posted 2012-04-16 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-03

CONDITIONS: Atopic Dermatitis; Eczema; Asthma; Food Allergies; Allergic Rhinitis
Keywords: Dermatitis; Eczema; Skin diseases; Skin barrier; Prevention; Infant; Moisturizer; Emollient; Asthma; Food allergy; Allergic rhinitis
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Asthma; Food Hypersensitivity; Rhinitis, Allergic; Dermatitis; Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: Lipikar Balm AP (Other): Daily application of Lipikar Balm AP starting at birth
  Interventions: Drug: Lipikar Balm AP
- Group 2: No intervention control group (No Intervention): Subjects may use a moisturizer if they wish to but no instruction or product is provided

INTERVENTIONS:
Drug: Lipikar Balm AP — Daily application of Lipikar Balm AP starting at birth
  Arms: Group 1: Lipikar Balm AP

SUMMARY:
There is a lack of prospective scientific data on the regular use of moisturizers in patients at risk of developing atopic dermatitis. Although generally accepted and widely used for secondary prevention, emollients have not been studied as a primary prevention strategy. Strategies previously studied for the prevention of atopic dermatitis include maternal and child's dietary manipulations, allergens avoidance, delay of food introduction, exclusive breastfeeding and probiotic supplementation. Despite years of research, none of those strategies yielded to strong evidence of a protective effect. There is therefore a need to explore novel strategies.

There is a need to compare the cumulative incidence rate of atopic dermatitis in newborns using a standard bathing and moisturizing routine with a good moisturizer to a non interventional group.

This 2-year study will recruit approximately four hundred and sixty (460) pregnant women with a first degree relative of the child to be born who currently has (or previously had) a diagnosis of atopic dermatitis in order to study approximately 200 eligible newborns in each of the two study groups at the beginning of the study.

Pregnant women will be randomized (1:1) to either daily use of the moisturizer Lipikar Balm AP (applied to their infant) starting from birth (Group 1) immediately after bathing or to no intervention (Group 2).

DETAILED DESCRIPTION:
To be eligible, pregnant women must be at least 16 weeks pregnant. Expecting mothers (or the father of the infant to be born) or related sibling of the child to be born must meet or previously have met criteria for atopic dermatitis. In addition, one of the parents or sibling of the child to be born must suffer from allergic rhinitis or asthma.

Pregnant women will be randomized at screening and their infant will be seen at 1 month, 6 months, 12 months (1 year) and 24 months (2 years) after birth.

Women randomized to group 1 will be requested to use the same body cleanser (Lipikar Syndet) and to apply Lipikar Balm AP to their child once daily immediately after bathing on a well blotted skin (within 3 minutes of bathing) to the entire body (including the face) from birth, while women randomized to group 2 will be in a non-interventional control group.

The presence of atopic dermatitis (using Hanifin's criteria(1)) and study products use will be assessed at 1 month, 6 months, 12 months and 24 months after birth. A buccal smear will be sampled from all infants at 1 month after birth for the genotyping of filaggrin (FLG) gene.

In addition, adverse events evaluation and parent questioning on infants development of food allergies and asthma will be performed at 1 month, 3 months (telephone visit), 6 months, 12 months and 24 months after birth. Infants will be followed for a total of two years after birth.

Lipikar Balm AP is a commonly used cosmetic moisturizer commercially available in many countries including Canada. This moisturizer is recommended for extreme dryness and atopy-prone skin in babies, children and adults. It contains shea butter, paraffin, waxes and vegetable oils. The high content in shea butter and the fraction chosen showed a greater expression of constitutive ceramids forming the barrier function of the skin (data on file at La Roche-Posay).

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older at the time of consent
* At least 16 weeks pregnant
* Women with a high risk of having a child with atopic dermatitis defined as having one parent or related sibling of the child to be born who currently (or previously) suffers from atopic dermatitis and who also suffers from asthma or allergic rhinitis
* Be willing to use the body cleanser Lipikar Syndet and to apply Lipikar Balm AP (if randomized to group 1) every day from birth for 2 years
* Capable of giving informed consent and the consent must be obtained prior to any study related procedures

Exclusion Criteria:

* Preterm birth defined as birth before 37 weeks of gestation
* Major congenital anomaly at birth
* Presence of significant dermatitis at birth
* Any medical problem at birth that would prevent the daily use of Lipikar Syndet and/or Lipikar Balm AP (regardless of the group the subject was randomized to) or would prevent evaluation of the skin for the presence of atopic dermatitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, FRCPC, Principal Investigator — Innovaderm Research
Locations (4):
- United States (2):
  - Hamzavi Dermatology/Dermatology Specialists of Canton, Canton, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
- Canada (2):
  - Lynderm Research, Markham, Ontario
  - Windsor Clinical Research, Windsor, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Screen Only: Subject was not randomized to either treatment prior to study termination.
Period: Overall Study
Arm/Group | Group 1: Lipikar Balm AP | Group 2: No Intervention Control Group | Screen Only
Started | 0 | 0 | 2
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Lipikar Balm AP | Group 2: No Intervention Control Group | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
Sex: Female, Male [Count of Participants; unit: Participants]
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Infants Who Develop Atopic Dermatitis
Description: Proportion of infants who develop atopic dermatitis at two years for infants randomized to Lipikar Balm AP as compared to infants randomized to the no intervention control group
Time Frame: 2 years
Population: Subjects were not randomized to either treatment prior to study termination and therefore no data was collected for this Outcome Measure
Arm/Group | Group 1: Lipikar Balm AP | Group 2: No Intervention Control Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Proportion of Infants Who Develop Asthma
Description: Proportion of infants who develop asthma at two years for infants randomized to Lipikar Balm AP as compared to infants randomized to the no intervention control group
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | Group 1: Lipikar Balm AP | Group 2: No Intervention Control Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Proportion of Infants Who Develop a Food Allergy
Description: Proportion of infants who develop a food allergy at two years for infants randomized to Lipikar Balm AP as compared to infants randomized to the no intervention control group
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | Group 1: Lipikar Balm AP | Group 2: No Intervention Control Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Influence of the Presence of Mutation in the Filaggrin Gene on the Proportion of Infants Who Develop Atopic Dermatitis
Description: Influence of the presence of mutation in the filaggrin gene on the proportion of infants who develop atopic dermatitis at two years for infants randomized to Lipikar Balm AP as compared to infants randomized to the no intervention control group
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | Group 1: Lipikar Balm AP | Group 2: No Intervention Control Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Influence of the Presence of Mutation in the Filaggrin Gene on the Proportion of Infants Who Develop Asthma
Description: Influence of the presence of mutation in the filaggrin gene on the proportion of infants who develop asthma at two years for infants randomized to Lipikar Balm AP as compared to infants randomized to the no intervention control group
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | Group 1: Lipikar Balm AP | Group 2: No Intervention Control Group
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Influence of the Presence of Mutation in the Filaggrin Gene on the Proportion of Infants Who Develop a Food Allergy
Description: Influence of the presence of mutation in the filaggrin gene on the proportion of infants who develop a food allergy at two years for infants randomized to Lipikar Balm AP as compared to infants randomized to the no intervention control group
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | Group 1: Lipikar Balm AP | Group 2: No Intervention Control Group
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Time of Onset of Asthma in Infants
Description: Time of onset of asthma in infants randomized to Lipikar Balm AP as compared to infants randomized to the no intervention control group
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | Group 1: Lipikar Balm AP | Group 2: No Intervention Control Group
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Time of Onset of Food Allergy in Infants
Description: Time of onset of food allergy in infants randomized to Lipikar Balm AP as compared to infants randomized to the no intervention control group
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | Group 1: Lipikar Balm AP | Group 2: No Intervention Control Group
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Adverse Events (AEs) Collection
Description: Adverse events (Skin AEs, asthma, food allergies, allergic rhinitis and any AE related to Lipikar Syndet, Lipikar Balm AP (group 1) or any other moisturizer application (group 2) will be collected.
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | Group 1: Lipikar Balm AP | Group 2: No Intervention Control Group
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Time of Onset of Atopic Dermatitis
Description: Time of onset of atopic dermatitis in infants randomized to Lipikar Balm AP as compared to infants randomized to the no intervention control group
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | Group 1: Lipikar Balm AP | Group 2: No Intervention Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The safety population is defined as all subjects who receive at least one dose of the study product until the end of study (2 years).
Description: Adverse events were only collected after subjects had their first dose of study product. Subjects were not randomized to either treatment prior to study termination and therefore no data was collected for Adverse Events. Adverse Events were not monitored/assessed for the two screened participants.
Arm/Group | Group 1: Lipikar Balm AP | Group 2: No Intervention Control Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No